CLINICAL TRIAL: NCT01958242
Title: The Effect of Preoperative Blood Harvesting and Its Re-administration at the End of Cardio-pulmonary Bypass on the Coagulation Profile in the Pediatric Population Undergoing Open Heart Surgery.
Brief Title: Effect of Blood Harvesting and Administration at End of CPB on Coagulation Profile
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical problems.
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 7192
Record Dates: First submitted 2013-04-17; First posted 2013-10-09 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2012-08

CONDITIONS: Hematologic Changes
Keywords: Cardiopulmonary bypass; pediatric; blood products; conservation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Preoperative blood harvesting (No Intervention)
  Interventions: Other: Preoperative blood harvesting

INTERVENTIONS:
Other: Preoperative blood harvesting — There is no true intervention, there is a protocol of preoperative blood harvesting ,and post operative administration of the same blood/

SUMMARY:
Blood transfusions after pediatric heart surgery is a relatively common practice occurring in up to 46% of patients, however its use has been associated with increased morbidity. In the pediatric population undergoing heart surgery transfusion of homologous blood is usually required due to the mismatch between the priming volume of the cardiopulmonary bypass circuit and the patients own blood volume. Several strategies have been proposed in order to minimize the use of blood products. The effect of pre-operative harvest of fresh whole blood in the adult population has shown a beneficial platelet protective effect, however concerns have been risen that the amount of volume needed in order to sequester a significant amount of platelets would be prohibit ally high in a cardiac surgical patient. Fresh blood harvesting has not been evaluated in the pediatric population.

The purpose of the present study would be to evaluate the safety and efficacy of pre-operative blood harvesting in the pediatric population undergoing open heart surgery. Fresh whole blood will be harvested from the patient prior to the initiation of cardiopulmonary bypass and will be returned to the patient after the discontinuation of CPB prior to the administration of prominent. Parameters that will be evaluated will include, patient characteristic, operative and post-operative parameters, coagulation profiles and the use of postoperative blood products.

DETAILED DESCRIPTION:
All pediatric patients undergoing open heart surgery at our institution will be randomized based on the last digit of their identification number (even or odd numbers) to undergo pre-operative whole blood harvesting (PBH). Informed consent will be obtained from the parents at the time of surgical informed consent acquisition.

After scrubbing and draping of the patient the first set of blood samples will be obtained for baseline.

Circuit priming will be performed using plasmalyte , and the prime will be adjusted to have a calculated bypass hematologic 27%, taking into consideration the amount of blood harvested.

Once the patient is connected to the CPB circuit, harvested blood will be taken from the venous line before its passage through the oxygenator, while crystalloids from the circuit will be infused through the arterial line in order to maintain adequate blood pressure. Once the amount of 15cc/kg of blood is harvested, CPB will be initiated and the operation will be carried out in the usual manner. Blood will be kept at room temperature (18°C), gently stirred (not shaken).

At the end of the operation, veno-venous ultrafiltration will be performed, targeting a duration of 10 minutes. The harvested blood will be administered at the end of ultrafiltration in conjunction to the administration of protamine. Blood samples will be obtained at various time points. Complete blood count, coagulation profile (PT/PTT), and platelet function tests will be performed. Pre-operative and operative characteristics will be recorded .

In the intensive care unit, the patient will be continuously followed until his discharge from the hospital and post-operative parameters will be recorded. Blood and blood product administration will be based on our ICU protocol and at the discretion of the attending physician. Generally, blood will be administered to single ventricle patients if their hemoglobin levels will be below 12 mg%, while in the 2 ventricle patients a threshold of 9mg% will be set. Administration of blood products will be performed if there will be signs of clinical bleeding with overt signs of coagulopathy (INR > 2, fibrinogen < 100, platelets < 50,000).

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients undergoing heart surgery

Exclusion Criteria:

* Unstable patients

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in coagulation profile | Immediate post operative
  Coagulation studies will be measured before and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Amir, MD, Principal Investigator — SCMCI
Locations (1):
- Schneider Children Medical center of Israel, Petah Tikva, Israel